CLINICAL TRIAL: NCT02199210
Title: Optimizing Intra-Operative Massive Transfusion: Probing for Forethought
Brief Title: Exploring Self-regulatory Processes in Anesthesiologists During Massive Transfusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Collaborators: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: SIMPROJECT-MT
Record Dates: First submitted 2014-07-21; First posted 2014-07-24 (Estimated); Last update posted 2016-08-10 (Estimated); Status verified 2016-08

CONDITIONS: Self-regulation; Forethought; Performance
Keywords: Massive transfusion protocols; Self-regulatory learning; Forethought; Clinical expertise; Simulation; Education
MeSH Terms: conditions — Self-Control

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prompting forethought (Experimental): A demographic questionnaire will be filled out by each participant. After randomization, participants will be presented with the background information of the simulated scenario.Subsequently:
  * participants forethought will be prompted and each participant will be asked to report his/her forethought,
  * participants then will be asked to manage a simulated massive transfusion scenario,
  * at completion of the scenario, each participant will undergo individualized debriefing and a syllabus on massive transfusion will be briefly discussed with them and also provided as a reading material for learning.
  Interventions: Other: Prompting forethought
- No prompting (No Intervention): A demographic questionnaire will be filled out by each participants. After randomization, participants will be presented with the background information of the simulated scenario.Subsequently:
  * participants will sit and wait for a predetermined time before entering into the simulator,
  * participants then will be asked to manage a simulated massive transfusion scenario,
  * at completion of the scenario, each participant will be interviewed about their thought process before entering to the simulation room,
  * each participant will undergo individualized debriefing and a syllabus on massive transfusion will be briefly discussed with them and also provided as a reading material for learning.

INTERVENTIONS:
Other: Prompting forethought — Participants will be asked questions which elicit specific forethought elements related to the given clinical situation. These are elements that relate to strategic planning, goal setting, goal orientation, imagery, outcome expectation. These context specific questions will be determined in the Pilot study and validated in Study I.
  Arms: Prompting forethought

SUMMARY:
The purpose of the project is to investigate the function of self-regulatory processes in anesthesiologists and how application of these processes influence performance in a crisis situation.The investigators intend to explore specifically the first phase of self-regulation, i.e. the forethought phase which describes processes related to strategic planning, goal setting, goal orientation, and outcome expectation. The investigators hypothesize that prompting forethought before engaging in a simulated massive transfusion crisis situation will result in better task performance in anesthesiologists.

DETAILED DESCRIPTION:
The investigators will conduct 3 studies building on each other.

* Pilot Study: the purpose of this study is to develop measurement tools for forethought, performance and a tool for prompting forethought. This study will include 2 attending anesthesiologists and 2 anesthesia residents (PGY2, 5).
* Study I: the purpose of this study is to validate the measurement tools for forethought, performance and the tool for prompting forethought. This will include 6 attending anesthesiologists, 6 PGY5 and 6 PGY2 anesthesia residents.
* Study II: the purpose of this study is to investigate if prompting forethought in anesthesia residents will result in better performance in a simulated massive transfusion than no prompting.

ELIGIBILITY:
Inclusion Criteria:

* Pilot study: attending anesthesiologists at St. Michael's Hospital , PGY5, PGY2 anesthesia residents at University of Toronto
* Study I: attending anesthesiologists at St. Michael's Hospital, PGY5, PGY2 anesthesia residents at University of Toronto
* Study II: PGY2, PGY3, PGY4 anesthesia residents at University of Toronto

Exclusion Criteria:

* Refusal to take part in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Performance in managing simulated massive transfusion scenario | Each individual's performance will be video recorded and subsequently evaluated within 8 weeks.
  Task specific performance tool will be developed in the Pilot study and will be validated in Study I. Each performance will be video recorded and two independent, blinded rater will evaluate the videos and assess performance. Performance assessment tool will be numerical including a 1-5 point scale for each performance element and a Global Rating Scale. Difference between massive transfusion management performance will be compared in anesthesia residents whose forethought is prompted to residents who don't receive prompting.

SECONDARY OUTCOMES:
Correlation between forethought scores and performance scores. | Forethought scores and performance scores will be determined within 8 weeks after individuals participated in the study.
  The investigators will determine if quality of forethought relates to quality of performance in anesthesia residents managing the simulated massive transfusion scenario. The Pilot study and Study I will be used to develop and validate a scoring form for forethought. This will include scores (1-5) for each forethought elements (strategic planning, goal setting, goal orientation, imaginary, outcome expectation) and a GRS (1-5).

OTHER OUTCOMES:
Development and validation of measurement tools for forethought, performance and a tool for prompting forethought. | Within 4 weeks after completion of Pilot study and Study I.
  In the Pilot study, think-aloud protocol will be used to identify forethought elements in experts (attending anesthesiologists) and non-expert (anesthesia residents). The real-time interviews will be used to design the measurement tool for forethought and also to develop a tool for prompting forethought. Equally, performance in a simulated massive transfusion scenario in experts and non-experts will be used to develop a scoring format for performance. The provisional scoring format then will be reviewed by experts and the research group. Study I will determine construct and predictive validity and reproducibility (inter-rater reliability) of these measurement scores.

CONTACTS AND LOCATIONS:
Overall Officials: John G Laffey, MD, FCARCSI, Principal Investigator — St. Michael's Hospital, University of Toronto; Charlotte Ringsted, PhD, Principal Investigator — The Wilson Center, University Health Network, University of Toronto
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Zimmermann BJ. Development of adaptation of expertise: The role of self-regulatory processes and beliefs. In: Ericsson KA, ed. The Cambridge Handbook of Expertise and Expert Performance: Cambridge Unicersity Press 2006:705-22.
- [Background] Ericsson KA. Protocol analysis and expert thought: concurrent verbalisations of thinking during experts' performance on representative tasks. In: Ericsson KA, ed. The Cambridge Handbook of Expertise and Expert Performance: Cambridge University Press 2006:223-41.
- [Background] Artino AR Jr, Cleary TJ, Dong T, Hemmer PA, Durning SJ. Exploring clinical reasoning in novices: a self-regulated learning microanalytic assessment approach. Med Educ. 2014 Mar;48(3):280-91. doi: 10.1111/medu.12303. PMID 24528463
- [Background] Cleary TJ, Sandars J. Assessing self-regulatory processes during clinical skill performance: a pilot study. Med Teach. 2011;33(7):e368-74. doi: 10.3109/0142159X.2011.577464. PMID 21696270
- [Background] Brydges R, Nair P, Ma I, Shanks D, Hatala R. Directed self-regulated learning versus instructor-regulated learning in simulation training. Med Educ. 2012 Jul;46(7):648-56. doi: 10.1111/j.1365-2923.2012.04268.x. PMID 22691145
- [Background] Dzik WH, Blajchman MA, Fergusson D, Hameed M, Henry B, Kirkpatrick AW, Korogyi T, Logsetty S, Skeate RC, Stanworth S, MacAdams C, Muirhead B. Clinical review: Canadian National Advisory Committee on Blood and Blood Products--Massive transfusion consensus conference 2011: report of the panel. Crit Care. 2011;15(6):242. doi: 10.1186/cc10498. Epub 2011 Dec 8. PMID 22188866
- [Background] Cotton BA, Dossett LA, Au BK, Nunez TC, Robertson AM, Young PP. Room for (performance) improvement: provider-related factors associated with poor outcomes in massive transfusion. J Trauma. 2009 Nov;67(5):1004-12. doi: 10.1097/TA.0b013e3181bcb2a8. PMID 19901661